CLINICAL TRIAL: NCT07397091
Title: ROUTINE INFLAMMATORY AND METABOLIC BIOMARKERS. Can They Predict a Positive Head CT in Paediatric Minor Traumatic Brain Injury?
Brief Title: Using Routine Inflammatory and Metabolic Blood Tests (Bedside Included) to Predict Brain Injury in Children After Minor Head Trauma
Acronym: paeds_mTBI_Bio
Status: Not yet recruiting | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Collaborators: Children's Emergency Clinical Hospital Cluj-Napoca (Unknown)
Responsible Party: Principal Investigator, Eugenia-Maria Lupan-Muresan, Associated Professor, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: DEP23/21.01.2026
Record Dates: First submitted 2026-01-30; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Brain Injury Traumatic Mild
Keywords: routine biomarkers; traumatic brain injury; inflammatory; metabolic
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 0 to 18, mild TBI (GCS 14-15 or A on AVPU): Patients aged 0 to 18 years old presenting to the ED with mild traumatic brain injury (with or without cervical injury):
  1. Mild TBI will be defined as GCS 14-15 or A (AVPU) upon admission
  2. Patients underwent head CT
  3. Routine blood biomarkers have been collected (complete blood count - CBC, biochemistry and/or (arterial) venos blood gases - (A)VBG).

SUMMARY:
Traumatic brain injury (TBI) poses significant strains on the paediatric population, for which the possible side effects of diagnostic imagistics could induce life-altering conditions. Routine inflammatory and metabolic biomarkers (complete blood count, C reactive protein, glucose) are frequently sampled in the paediatric patients admited within emergency departments, including the low-resource settings. This study aims to retrospectively document whether such routine blood biomarkers could predict a positive head CT scan and subsequently contribute to a prediction score, ment to enable more accurate decision on which minor TBI paediatric patients should be submitted to diagnotic imagistics.

DETAILED DESCRIPTION:
Epidemiology and Clinical Context Traumatic brain injury (TBI) is a significant global health concern, with an estimated paediatric global annual incidence of 226.4 cases per 100,000 children (1). The vast majority of these cases are categorized as non-severe, as up to 95% of head injuries in children are classified as minor or mild (mTBI) (1,2). Nevertheless, approximately one-third of paediatric patients experience persistent symptoms lasting beyond one month (3).

The current diagnostic gold standard remains non-contrast head Computed Tomography (CT). However, CT utilization carries significant associated risks, including exposure to ionizing radiation, high institutional costs, and the frequent necessity for procedural sedation (4). To mitigate these risks, clinical decision rules such as PECARN, CATCH, and CHALICE were developed to identify children at high risk for intracranial lesions. Despite these tools, most CT scans are still performed in cases of mTBI where the diagnostic yield is remarkably low (5).

As such, additional aiding tools have been investigated for refining the clinical decision rules regarding the paediatric mTBI patients in need of a CT scan.

Brain-Specific Biomarkers (GFAP, UCH-L1, S100B) In 2018, the US FDA authorized the first biomarkers (GFAP and UCH-L1) for predicting the necessity of CT scans in patients with minor TBI, supported by the ALERT-TBI trial (6). These markers serve as critical tools for both diagnosis and prognosis in neurotrauma (7).

GFAP (Glial Fibrillary Acidic Protein) is an astroglial protein that can predict positive CT findings in children with a sensitivity of 94% and a specificity of 47% (8). Its high sensitivity makes it an ideal "rule-out" marker.

UCH-L1 (Ubiquitin C-terminal Hydrolase L1) is a neuronal marker released into the bloodstream following axonal injury (6).

While extensively studied, S100B has shown limitations in paediatric emergency care. Research by Babcock et al. (2012) demonstrated it could not accurately predict positive CT findings in children with a normal GCS (9). Furthermore, its specificity is hindered by age-dependent baseline levels (10).

Routine Hematological and Metabolic Markers Beyond brain-specific proteins, routine complete blood count (CBC) parameters and metabolic markers provide an immediate, cost-effective snapshot of the injury's systemic impact, additionally to being easily accessible even in low-resource environments.

1. Inflammatory Indexes (NLR, Delta NLR, SII) Paediatric TBI patients with intracranial lesions on imaging demonstrate a significantly higher absolute neutrophil count (11).

   Significant differences in the Neutrophil-to-Lymphocyte Ratio (NLR) are observed at 24 and 48 hours post-injury (12,13). Longitudinal changes (Delta NLR) are associated with poorer clinical outcomes in children (14).

   The Systemic Immune-Inflammation Index (SII) (Neutrophils × Platelets / Lymphocytes) is increasingly used to monitor the secondary inflammatory cascade (15).
2. Glucose as a Modifiable Risk Factor Metabolic distress, specifically hyperglycemia, is a critical factor in the acute phase of TBI.

Admission glucose levels are a potentially modifiable risk factor in TBI; elevated glucose is closely linked to the severity of the primary injury (16) and the occurrence of coagulopathy in TBI patients, further complicating the clinical trajectory (17). Elevated blood glucose levels may aid clinicians in the decision-making process for ordering CT scans in cases of minor head trauma (18).

Conclusion The integration of specialized biomarkers like GFAP and UCH-L1 offers high sensitivity for ruling out acute pathology, yet their availability remains limited in the setting of emergency care. As such, routine biomakers, such as glucose levels, CBC panel and its derived inflammatory indexes, could provide relevant prognostic data in a more cost-effective approach for the triage and monitoring of emergency department paediatric mTBI, whilst limiting the radiation exposure of paediatric patients.

References

1. Baticulon RE, Sy JJ, Haizel-Cobbina J, et al. Global Epidemiology of Pediatric Traumatic Brain Injury: Systematic Review and Meta-Analysis. Neurosurgery. 2025. doi: 10.1227/neu.0000000000003875. Epub ahead of print. PMID: 41384742.
2. Babl FE, Borland ML, Phillips N, et al. Accuracy of PECARN, CATCH, and CHALICE decisions rules for children with minor head injury: a prospective cohort study. Lancet. 2017;389(10087):2393-402.
3. Eisenberg MA, Andrea J, Meehan W, Mannix R . Time interval between concussions and symptom duration. Pediatrics. 2013;132(1):8-17. PMID: 23753087. DOI: 10.1542/peds.2013-0432.
4. Sheppard JP, Nguyen T, Alkhalid Y, et al. Risk of Brain Tumor Induction from Pediatric Head CT Procedures: A Systematic Literature Review. J Pediatr Surg. 2018;53(12):2450-2455. DOI:10.1016/j.jpedsurg.2018.04.032.
5. Marincowitz C, Lecky FE, Townend W, et al. The Risk of Deterioration in GCS13-15 Patients with Traumatic Brain Injury Identified by Computed Tomography Imaging: A Systematic Review and Meta-Analysis. J Neurotrauma. 2018; 35(5):703-718. PMID: 29324173. DOI: 10.1089/neu.2017.5259.
6. Bazarian JJ, Biberthaler P, Welch RD, et al. Serum GFAP and UCH-L1 for prediction of absence of intracranial injuries on head CT (ALERT-TBI): a multicentre observational study. Lancet Neurol. 2018;17(9):782-789. PMID: 30054151. Doi: 10.1016/S1474-4422(18)30231-X.
7. Wang KK, Yang Z, Zhu T, et al. An update on diagnostic and prognostic biomarkers for traumatic brain injury. Expert Rev Mol Diagn. 2018;18(2):165-180. PMID: 29338452. DOI: 10.1080/14737159.2018.1428089.
8. Papa L, Brophy GM, Welch RD, et al. Time Course and Diagnostic Accuracy of Glial and Neuronal Blood Biomarkers GFAP and UCH-L1 in a Large Cohort of Trauma Patients With and Without Mild Traumatic Brain Injury. JAMA Neurol. 2016;73(5):551-60. PMID: 27018834. DOI: 10.1001/jamaneurol.2016.0039.
9. Babcock L, Byczkowski T, Mookerjee S, Bazarian JJ. Ability of S100B to predict severity and cranial CT results in children with TBI. Brain Inj. 2012;26(11):1372-80. PMID: 22725661. DOI: 10.3109/02699052.2012.694565.
10. Oris C, Pereira B, Durif J, et al. The Biomarker S100B and Mild Traumatic Brain Injury: A Meta-analysis. Pediatrics. 2018;141(6):e20180037. PMID: 29716980. DOi: 10.1542/peds.2018-0037.
11. Mukherjee S, Sivakumar G, Goodden JR, Tyagi AK, Chumas PD. Prognostic value of leukocytosis in pediatric traumatic brain injury. J Neurosurg Pediatr. 2020;27(3):335-345. PMID: 33361484. DOI: 10.3171/2020.7.PEDS19627..
12. Siempis T, Georgalis PA, Lianos G, et al. Blood Biomarkers for Prediction of Positive CT Findings in Mild Traumatic Brain Injury in Paediatric Population. J Integr Neurosci. 2023;22(4):91. PMID: 37519178. DOI: 10.31083/j.jin2204091.
13. Kimball R, Shachar E, Eyerly-Webb S, Patel DM, Spader H. Using the neutrophil-to-lymphocyte ratio to predict outcomes in pediatric patients with traumatic brain injury. Clin Neurol Neurosurg. 2020;193:105772. PMID: 32155528. DOI: 10.1016/j.clineuro.2020.105772.
14. Melo JRT, Masini MHH, de Oliveira JG, Veiga JCE. Performance of the neutrophil-lymphocyte ratio as a predictor of severity and mortality in children and adolescents with traumatic brain injury. Childs Nerv Syst. 2024;40(12):4251-4257. PMID: 39080015. DOI: 10.1007/s00381-024-06556-9.
15. Parenrengi MA, Suryaningtyas W, Dariansyah AD, Utomo B, Taryana GO, Kusumo C, et al. Utility of systemic immune-inflammation index, neutrophil-to-lymphocyte ratio, and platelet-to-lymphocyte ratio as a predictive biomarker in pediatric traumatic brain injury. Surg Neurol Int. 2024;15:456. PMID: 39777169. DOI: 10.25259/SNI_900_2024.
16. Shi J, Dong B, Mao Y, et al. Review: traumatic brain injury and hyperglycemia, a potentially modifiable risk factor. Oncotarget. 2016;7(43):71052-71061. PMID: 27626493.
17. Alexiou GA, Lianos G, Fotakopoulos G, et al. Admission glucose and coagulopathy occurrence in patients with traumatic brain injury. Brain Inj. 2014;28(4):438-441. PMID: 24564221.
18. Alexiou GA, Sotiropoulos A, Lianos GD, et al. Blood Glucose levels may aid the decision for CT scan in minor head trauma. Dis Markers. 2019;2019:1065254. PMID: 31093304.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 0 to 18 years old presenting to the ED with mild traumatic brain injury (with or without cervical injury):

1. Mild TBI will be defined as GCS 14-15 or A (AVPU) upon admission
2. Patients underwent head CT
3. Routine blood biomarkers have been collected (complete blood count - CBC, biochemistry and/or (arterial) venos blood gases - (A)VBG).

Exclusion Criteria:

* Patients with moderate (GCS 13-9 or V) or severe (GCS 8-3 or P,U) head trauma
* Patients with associated trauma (limb/rib/pelvic fractures, organ injuries).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric patients being admitted to ED for minor traumatic brain injuries, who are undergoing a head CT scan and routine blood tests.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2026-04-20 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Routine Biomarkers | Upon ED admission for mTBI
  1. CBC, the following items being mandatory:
     * WBC (white blood cells) and its subpopulations (NEU, LYM, MON)
     * NLR (neutrophiles-to-lymphocytes ratio)
     * PLR (platelets-to-lymphocyes ratio)
     * MLR (monocytes-to-lymphocytes ratio)
     * SII (systemic immune inflammation) index = NEU x PLT/ LYM
     * SIRI (systemic inflammatory response index) = NEU x MON/ LYM
  2. C Reactive Protein
  3. Glucose
  4. (A)VBG - pH, lactate, base deficit, anion gap, bicarb

SECONDARY OUTCOMES:
Epidemiological Data | Upon ED admission for mTBI
  Additionally, epidemological data will be collected (age, gender, trauma mechanism, associated lessions, risk factors for TBI classification, physical examination, need of procedural sedation, seniority of treating physician, disposition), alongside the results of the head (and cervical) CT scan.

OTHER OUTCOMES:
TBI Registry | Upon ED admission for mTBI
  A TBI registry will be also filled in, registering all TBI patients who do not meet the study inclusion criteria (mTBI without CT scan, moderate and severe TBI). For these patients, the collected data are the following:
  * patient ID
  * gender, age
  * GCS upon admission
  * TBI severity (as mentioned in the final ED diagnosis)
  * seniority of treating physician

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia M Lupan-Muresan, MD, PhD, Principal Investigator — Iuliu Hatieganu University of Medicine and Pharmacy Cluj-Napoca; Daniela M Mitrofan, MD, Principal Investigator — Children's Emergency County Hospital Cluj-Napoca
Locations (7):
- Romania (7):
  - Spitalul Clinic Judetean de Urgenta, Arad
  - Spitalul Judetean de Urgenta, Baia Mare
  - Spitalul Clinic Judetean de Urgenta, Bistriţa
  - Spitalul Judetean de Urgenta MAVROMATI, Botoșani
  - Spitalul Clinic de Urgenta penru Copii, Brasov
  - Spitalul Clinic de Urgenta pentru Copii, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta, Craiova

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alexiou GA, Sotiropoulos A, Lianos GD, Zigouris A, Metaxas D, Nasios A, Michos E, Mitsis M, Pachatouridis D, Voulgaris S. Blood Glucose Levels May Aid the Decision for CT Scan in Minor Head Trauma. Dis Markers. 2019 Apr 9;2019:1065254. doi: 10.1155/2019/1065254. eCollection 2019. PMID 31093304
- [Background] Alexiou GA, Lianos G, Fotakopoulos G, Michos E, Pachatouridis D, Voulgaris S. Admission glucose and coagulopathy occurrence in patients with traumatic brain injury. Brain Inj. 2014;28(4):438-41. doi: 10.3109/02699052.2014.888769. Epub 2014 Feb 24. PMID 24564221
- [Background] Shi J, Dong B, Mao Y, Guan W, Cao J, Zhu R, Wang S. Review: Traumatic brain injury and hyperglycemia, a potentially modifiable risk factor. Oncotarget. 2016 Oct 25;7(43):71052-71061. doi: 10.18632/oncotarget.11958. PMID 27626493
- [Background] Parenrengi MA, Suryaningtyas W, Dariansyah AD, Utomo B, Taryana GO, Kusumo C, Brilliantika SP. Utility of systemic immune-inflammation index, neutrophil-to-lymphocyte ratio, and platelet-to-lymphocyte ratio as a predictive biomarker in pediatric traumatic brain injury. Surg Neurol Int. 2024 Dec 6;15:456. doi: 10.25259/SNI_900_2024. eCollection 2024. PMID 39777169
- [Background] Melo JRT, Masini MHH, de Oliveira JG, Veiga JCE. Performance of the neutrophil-lymphocyte ratio as a predictor of severity and mortality in children and adolescents with traumatic brain injury. Childs Nerv Syst. 2024 Dec;40(12):4251-4257. doi: 10.1007/s00381-024-06556-9. Epub 2024 Jul 30. PMID 39080015
- [Background] Mukherjee S, Sivakumar G, Goodden JR, Tyagi AK, Chumas PD. Prognostic value of leukocytosis in pediatric traumatic brain injury. J Neurosurg Pediatr. 2020 Dec 25;27(3):335-345. doi: 10.3171/2020.7.PEDS19627. Print 2021 Mar 1. PMID 33361484
- [Background] Kimball R, Shachar E, Eyerly-Webb S, Patel DM, Spader H. Using the neutrophil-to-lymphocyte ratio to predict outcomes in pediatric patients with traumatic brain injury. Clin Neurol Neurosurg. 2020 Jun;193:105772. doi: 10.1016/j.clineuro.2020.105772. Epub 2020 Mar 3. PMID 32155528
- [Background] Siempis T, Georgalis PA, Lianos G, Kafritsas G, Metaxas D, Alexiou ES, Zika J, Sotiropoulos A, Alexiou GA, Voulgaris S. Blood Biomarkers for Prediction of Positive CT Findings in Mild Traumatic Brain Injury in Paediatric Population. J Integr Neurosci. 2023 Jul 7;22(4):91. doi: 10.31083/j.jin2204091. PMID 37519178
- [Background] Oris C, Pereira B, Durif J, Simon-Pimmel J, Castellani C, Manzano S, Sapin V, Bouvier D. The Biomarker S100B and Mild Traumatic Brain Injury: A Meta-analysis. Pediatrics. 2018 Jun;141(6):e20180037. doi: 10.1542/peds.2018-0037. Epub 2018 May 1. PMID 29716980
- [Background] Babcock L, Byczkowski T, Mookerjee S, Bazarian JJ. Ability of S100B to predict severity and cranial CT results in children with TBI. Brain Inj. 2012;26(11):1372-80. doi: 10.3109/02699052.2012.694565. Epub 2012 Jun 22. PMID 22725661
- [Background] Papa L, Brophy GM, Welch RD, Lewis LM, Braga CF, Tan CN, Ameli NJ, Lopez MA, Haeussler CA, Mendez Giordano DI, Silvestri S, Giordano P, Weber KD, Hill-Pryor C, Hack DC. Time Course and Diagnostic Accuracy of Glial and Neuronal Blood Biomarkers GFAP and UCH-L1 in a Large Cohort of Trauma Patients With and Without Mild Traumatic Brain Injury. JAMA Neurol. 2016 May 1;73(5):551-60. doi: 10.1001/jamaneurol.2016.0039. PMID 27018834
- [Background] Wang KK, Yang Z, Zhu T, Shi Y, Rubenstein R, Tyndall JA, Manley GT. An update on diagnostic and prognostic biomarkers for traumatic brain injury. Expert Rev Mol Diagn. 2018 Feb;18(2):165-180. doi: 10.1080/14737159.2018.1428089. Epub 2018 Jan 23. PMID 29338452
- [Background] Bazarian JJ, Biberthaler P, Welch RD, Lewis LM, Barzo P, Bogner-Flatz V, Gunnar Brolinson P, Buki A, Chen JY, Christenson RH, Hack D, Huff JS, Johar S, Jordan JD, Leidel BA, Lindner T, Ludington E, Okonkwo DO, Ornato J, Peacock WF, Schmidt K, Tyndall JA, Vossough A, Jagoda AS. Serum GFAP and UCH-L1 for prediction of absence of intracranial injuries on head CT (ALERT-TBI): a multicentre observational study. Lancet Neurol. 2018 Sep;17(9):782-789. doi: 10.1016/S1474-4422(18)30231-X. Epub 2018 Jul 24. PMID 30054151
- [Background] Marincowitz C, Lecky FE, Townend W, Borakati A, Fabbri A, Sheldon TA. The Risk of Deterioration in GCS13-15 Patients with Traumatic Brain Injury Identified by Computed Tomography Imaging: A Systematic Review and Meta-Analysis. J Neurotrauma. 2018 Mar 1;35(5):703-718. doi: 10.1089/neu.2017.5259. Epub 2018 Jan 11. PMID 29324173
- [Background] Sheppard JP, Nguyen T, Alkhalid Y, Beckett JS, Salamon N, Yang I. Risk of Brain Tumor Induction from Pediatric Head CT Procedures: A Systematic Literature Review. Brain Tumor Res Treat. 2018 Apr;6(1):1-7. doi: 10.14791/btrt.2018.6.e4. PMID 29717567
- [Background] Eisenberg MA, Andrea J, Meehan W, Mannix R. Time interval between concussions and symptom duration. Pediatrics. 2013 Jul;132(1):8-17. doi: 10.1542/peds.2013-0432. Epub 2013 Jun 10. PMID 23753087
- [Background] Babl FE, Borland ML, Phillips N, Kochar A, Dalton S, McCaskill M, Cheek JA, Gilhotra Y, Furyk J, Neutze J, Lyttle MD, Bressan S, Donath S, Molesworth C, Jachno K, Ward B, Williams A, Baylis A, Crowe L, Oakley E, Dalziel SR; Paediatric Research in Emergency Departments International Collaborative (PREDICT). Accuracy of PECARN, CATCH, and CHALICE head injury decision rules in children: a prospective cohort study. Lancet. 2017 Jun 17;389(10087):2393-2402. doi: 10.1016/S0140-6736(17)30555-X. Epub 2017 Apr 11. PMID 28410792
- [Background] Baticulon RE, Sy JJ, Haizel-Cobbina J, Du L, Figueredo L, Hounjet C, Mitchell R, Shlobin NA, Dewan MC. Global Epidemiology of Pediatric Traumatic Brain Injury: Systematic Review and Meta-Analysis. Neurosurgery. 2025 Dec 12. doi: 10.1227/neu.0000000000003875. Online ahead of print. PMID 41384742